CLINICAL TRIAL: NCT00933049
Title: Clinical Efficacy of Cotrimoxazole Versus Amoxicillin in the Treatment of Community Acquired Pneumonia in Children Aged 2-59 Months Attending Mulago Hospital: A Randomized Clinical Trial.
Brief Title: Cotrimoxazole Versus Amoxicillin in the Treatment of Community Acquired Pneumonia in Children Aged 2-59 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Prof James K Tumwine, Faculty of Medicine, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005HD11/3472U
Record Dates: First submitted 2009-07-05; First posted 2009-07-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Childhood Pneumonia
Keywords: Efficacy; children; pneumonia; cotrimoxazole; amoxicillin
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cotrimoxazole (Active Comparator): Cotrimoxazole (8 mg/kg/dose trimethoprim + 40 mg/kg/dose sulphamethoxazole) + Amoxicillin placebo
  Interventions: Drug: Cotrimoxazole; Drug: Amoxicillin placebo
- Amoxicillin (Active Comparator): Amoxicillin (25 mg/kg/dose) + Cotrimoxazole placebo
  Interventions: Drug: Amoxicillin; Drug: Cotrimoxazole placebo

INTERVENTIONS:
Drug: Amoxicillin — Oral amoxicillin (25mg/kg/dose)for 5 days
  Other Names: AMOX
  Arms: Amoxicillin
Drug: Cotrimoxazole — Cotrimoxazole (8 mg/kg/dose trimethoprim + 40 mg/kg/dose sulphamethoxazole)
  Other Names: CTX
  Arms: Cotrimoxazole
Drug: Amoxicillin placebo
  Arms: Cotrimoxazole
Drug: Cotrimoxazole placebo
  Arms: Amoxicillin

SUMMARY:
The investigators hypothesized that Oral amoxicillin (25mg/kg/dose bid) given to children aged 2-59 months with pneumonia, would lead to better clinical outcome on day three in 89.9% of the children compared to 77.0% of children receiving oral cotrimoxazole (8 mg/kg/dose trimethoprim, 40 mg/kg/dose sulphamethoxazole). A double blind randomized controlled trial was conducted in the Assessment Center of Mulago Hospital. Children with non-severe pneumonia were randomized to receive either oral amoxicillin (25 mg/kg/dose) or cotrimoxazole (trimethoprim 8 mg/kg and sulphamethoxazole 40 mg/kg) and followed up on day 3 and 5 of treatment. The primary outcome measures were normalization of respiratory rate by day 3 of treatment. Secondary outcome measures were antimicrobial susceptibility to cotrimoxazole and amoxicillin.

DETAILED DESCRIPTION:
A triage Nurse identified and recorded children aged 2- 59 months who presented with a history of cough, difficult breathing, or fast breathing (tachypnea) in the Assessment Center of Mulago Hospital. Children aged 2-11 months with a respiratory rate>50 breaths per minute and those aged 12-59 months with a respiratory rate of > 40 breaths per minute were enrolled into the study following informed consent from parents/caretakers. Clinical history included the patient's detailed record of the illness, previous medical history and antibiotic use in the current illness. The IMCI approach was particularly employed during history taking and examination. The Principle Investigator and the research assistant interviewed the caretakers using a structured questionnaire. 5 mls of blood was drawn from the ante cubital fossa for a complete blood count and blood cultures.In addition thin and thick blood smears for malaria parasites were taken using finger prick blood samples. Rapid HIV antibody test was done to determine the HIV serostatus of the children. Children less than 18 months with a positive antibody test were referred to the Paediatric Infectious Disease Clinic (PIDC) Mulago Hospital for a DNA-PCR test to confirm their HIV infection status. Study participants were placed in a well aerated room and subjected to sputum induction. The principal investigator, with the help of the research assistant and a nurse performed the procedure.

The study patients were nebulised with salbutamol at a dose of 0.1mg/kg in 3ml of Normal saline. 3mls of 3% sterile saline was administered through a facemask nebuliser for about 10-15 minutes.Sputum was obtained by expectoration (in children who could do it) or by nasopharyngeal suction in those who were unable to expectorate. Gram stain, ZN stain and culture and sensitivity was performed on sputum. Oxygen saturation was measured before and after sputum induction. For those children who had oxygen saturation of less than 92% or could not tolerate the sputum induction, the procedure was deferred to the following day when the children were more stable. However, they continued with treatment. Treatment assignment was concealed from patients, parents, and study personnel. Children assigned co-trimoxazole received active medicine (8 mg/kg/dose trimethoprim + 40 mg/kg/dose sulphamethoxazole) and amoxicillin placebo twice a day. Children assigned amoxicillin received active medicine (25 mg/kg/dose) and co-trimoxazole placebo twice a day.A randomization scheme was developed using a table of random numbers generated by computer. Study participants were randomly assigned to treatment in blocks of 4 to 12. Both drugs and placebo were manufactured and packaged in volumes of 100mls and had the same color. Treatment was started as soon as patients were enrolled in the study after withdrawal of blood and sputum samples. Drug doses were calculated according to the body weight. Cotrimoxazole was given orally (syrup) in a dose of 8mg/kg/dose trimethoprim, 40mg/kg/dose sulphamethoxazole and oral (syrup) amoxicillin in a dose of 25mg/kg/dose every 12 hours until a total of 5 days was reached. The study had two treatment arms; one arm was randomly assigned to receive active amoxicillin plus placebo cotrimoxazole orally and the other arm was randomly assigned to receive active cotrimoxazole with placebo amoxicillin two doses per day. The study nurse and the principle investigator demonstrated to the parent/caretaker how to give the study drugs by giving the first dose from the clinic. An explanation was given on how to give medication at home and the level of understanding was checked before leaving clinic. Caretakers were instructed not to give any other medications especially antibiotics other than those given in the hospital and were instructed to return to the clinic on day 3 and 5 of treatment. Paracetamol syrup was administered to febrile children at a dose of 15 mg/kg 4 - 6 hourly if their axillary temperature were 38.5 degrees Celsius and above. Vitamin A was given according to the national recommendation guidelines. Patients who were diagnosed with malaria from blood slides were given Arthemeter-Lumefantrine tablets. Other medications were as well given according to the presentation and the diagnosis.The day of enrollment was counted as day 0. After three days of treatment, patients were checked for general danger signs and assessed for cough or difficult breathing and the respiratory rate counted. Improvement was defined as slower respiratory rate (either back to normal range for age, or more than 5 breaths per minute lower compared to the previous evaluation), less fever, normal oxygen saturation and better appetite, then patients were requested to complete the 5 days antibiotics and final follow up on the day 5 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-59 months with non severe pneumonia based on WHO criteria of respiratory rate above the age specific cut-off
* Accessible to follow up
* Written informed consent from the parent/caretaker

Exclusion Criteria:

* Children with severe pneumonia
* Documented use of antibiotics for the last 48 hours
* Confirmed HIV positive on cotrimoxazole prophylaxis
* Three or more episodes of wheezing in a year with asthmatic attack
* History of hospitalization within last 15 days
* Measles within last one month
* Previous history of allergy to cotrimoxazole or amoxicillin

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 505 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Normalisation of respiratory rate to age specific range by day 3 of treatment | 3 days

SECONDARY OUTCOMES:
Antimicrobial susceptibility to cotrimoxazole and amoxicillin | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Joyce M Kaducu, MBChB, MMED, Principal Investigator — Makerere University
Locations (1):
- Faculty of Medicine, Makerere University, Kampala, Uganda